CLINICAL TRIAL: NCT04502186
Title: A Systems-Level Intervention for Rural Adults With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Addie Weaver, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00176192; K01MH110605 (NIH)
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raising Our Spirits Together Intervention (Experimental)
  Interventions: Behavioral: Raising Our Spirits Together
- Enhanced Control Condition (Other)
  Interventions: Other: Enhanced Control Condition

INTERVENTIONS:
Behavioral: Raising Our Spirits Together — Raising Our Spirits Together (ROST) is an 8-session computer-assisted cognitive behavioral therapy for depression. Core CBT content, including behavioral activation, cognitive restructuring, and problem solving, are delivered via the computer-assisted platform using video and text-based elements. The computer-assisted intervention is complemented by a workbook that includes in-session exercises as well as homework/action plans. ROST is delivered weekly, either virtually or in-person at a local church, and facilitated by a local pastor.
  Arms: Raising Our Spirits Together Intervention
Other: Enhanced Control Condition — The Enhanced Control Condition intervention consists of providing participants randomized to this condition with a self-help book for depression (The Depression Helpbook; Katon et al, 2008) that is widely used and found to be beneficial, a local resource guide, and referrals.
  Arms: Enhanced Control Condition

SUMMARY:
This study aims to test the effectiveness of a computer-assisted cognitive behavioral therapy for depression among rural adults. The intervention, called Raising Our Spirits Together (ROST), was developed via a community-based participatory approach and will be delivered in small groups, facilitated by local pastors. Groups will be held virtually, or in-person at two churches in rural Michigan. Eighty-four individuals will be recruited from Hillsdale, Michigan, to test the effect of ROST on depressive symptoms, compared to an Enhanced Control Condition (ECC).

ELIGIBILITY:
Inclusion Criteria:

* Must live in Hillsdale, Lenawee, Jackson, or Calhoun County, Michigan
* Positive screen for at least mild depressive symptoms based on the the Patient Health Questionnaire-9 (PHQ-9>=5)

Exclusion Criteria:

* Non-English speaking
* Currently receiving cognitive behavioral therapy (CBT) for depression
* Ever completed a course of cognitive behavioral therapy (CBT; >=8 sessions)
* Diagnosis of a psychotic disorder
* Current use of opiates or freebase cocaine
* Prominent suicidal/homicidal ideation with imminent risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Addie Weaver, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Trinity Lutheran Church, Hillsdale, Michigan
  - Jonesville First Presbyterian Church, Jonesville, Michigan

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available through NIMH Data Archive (NDAR) after the end of the study.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Raising Our Spirits Together Intervention | Enhanced Control Condition
Started | 40 | 30
Completed | 29 | 20
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Raising Our Spirits Together Intervention: Raising Our Spirits Together (ROST) is an 8-session computer-assisted cognitive behavioral therapy for depression. Core CBT content, including behavioral activation, cognitive restructuring, and problem solving, are delivered via the computer-assisted platform using video and text-based elements. The computer-assisted intervention is complemented by a workbook that includes in-session exercises as well as homework/action plans. ROST is delivered weekly, either virtually or in-person at a local church, and facilitated by a local pastor.
- Total: Total of all reporting groups
Arm/Group | Raising Our Spirits Together Intervention | Enhanced Control Condition | Total
Number analyzed (Participants) | 40 | 30 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.63 (15.26) | 39.57 (13.68) | 43.03 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 9 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 39 | 27 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 3 | 7
  White | 35 | 25 | 60
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 30 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-report Measure of Depressive Symptoms
Description: Participants will self report depressive symptoms utilizing the Patient Health Questionnaire-9 (PHQ-9; range 0-27 with higher scores indicating worse outcome)
Time Frame: Outcome will be assessed at baseline, immediately post-treatment (up to 8 weeks), and 12-weeks post-treatment
Measure: Mean (Standard Deviation); unit: score on PHQ-9
Arm/Group | Raising Our Spirits Together Intervention | Enhanced Control Condition
Number analyzed (Participants) | 40 | 30
score on PHQ-9
  PHQ-9 Baseline | 13.90 (5.49) | 13.43 (4.40)
  PHQ-9 Post-treatment | 7.00 (5.67) | 7.57 (4.03)
  PHQ-9 Follow-up | 7.72 (7.36) | 8.10 (5.51)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant from the time of enrollment through study completion, which was, on average, 6 months.
Arm/Group | Raising Our Spirits Together Intervention | Enhanced Control Condition
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/30
Other Adverse Events (participants affected / at risk) | 1/40 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raising Our Spirits Together Intervention (N=40) | Enhanced Control Condition (N=30)
Protocol Deviation (Social circumstances) | 1 (1) | 0 (0) — A research associate mailed one participant's research incentive check to the wrong address. It was mailed to another research participant's home.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT04502186/Prot_SAP_000.pdf